CLINICAL TRIAL: NCT04386382
Title: Evaluation of Interchangeable Guide in Flapless Ridge Splitting With Simultaneous Implant Placement (Clinical Study)
Brief Title: Interchangeable Guide in Ridge Splitting Flapless Technique for Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ridge splitting
Record Dates: First submitted 2020-05-07; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Anterior Maxillary Narrow Ridge

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ridge splitting flapless technique using interchangeable guide (Experimental): Fabrication of interchangeable surgical guide stent:
  * Optical scanning of the dental casts was done using Ceramill map 400
  * The treatment plan and the surgical stent were designed using Mimics Innovation Suite 19 ™ software
  * Series of creating and designing special 3D virtual guide slits and boxes that can accommodate and precisely fit the tools used for the ridge splitting technique.
  Interventions: Procedure: ridge splitting flapless technique using interchangeable guide followed by implant placement

INTERVENTIONS:
Procedure: ridge splitting flapless technique using interchangeable guide followed by implant placement — An informed consent is taken from all the patients
  I. Presurgical phase:
  1. Proper dental and medical history.
  2. Scaling and oral hygiene measurements.
  3. Clinical examination.
  4. Radiographic examination. Clinical bucco-lingual measurements was done using calipers to ensure the patients would meet our initial inclusion criteria prior to further investigations.
  III. Fabrication of interchangeable surgical guide stent from primary impression:
  1. Optical scanning of the dental casts was done using Ceramill map 400
  2. surgical stent was designed using Mimics Innovation Suite 19 ™ software.
  3. Series of creating and designing special 3D virtual guide slits and boxes that can accommodate and precisely fit the tools used for the ridge splitting technique.
  All patients will be operated under local anesthesia, stent was placed on ridge and adapted well after disinfection osteotomy was done using piezotome splitting tips Implant-insertion was started immediately

SUMMARY:
A clinical trial was conducted to evaluate the accuracy of dental implant placement in narrow ridges after ridge splitting flapless technique using an interchangeable guide.

DETAILED DESCRIPTION:
A sample was selected conveniently to fulfill a list of inclusion and exclusion criteria. Then the selected participants underwent ridge splitting with the aid of interchangeable guide. After ridge splitting, all patients had simultaneous implant placement followed by clinical and radiographical evaluation over a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anterior maxillary narrow ridge
* Patients with adequate alveolar ridge bone height
* Age ranging from 20-40 years.
* Patients should have adequate oral hygiene
* Patients should be free of soft tissue or oral dental pathology
* Patients who accept to participate in the study.

Exclusion Criteria:

* Patients suffering from relevant systemic and/or metabolic diseases
* Patients suffering from immunosuppressive and/or autoimmune diseases
* Heavy smokers.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Clinical evaluaion | After 1 week
  post operative complication (presence or absence of any sign of swelling or infection)
Postoperative Pain | After 1 week
  Visual Analouge Scale (VAS) 0=no pain
  1. mild pain; it is easily tolerated
  2. moderate pain; it is causing discomfort but bearable.
  3. severe pain; it is causing discomfort, hardly tolerated and unbearable.
Change of bone width from baseline measurements | Baseline, 1 week, 3 months and 6 months
  Cone beam computed tomography (CBCT) was used to evaluate bone width and density to all patients by doing CBCT at time intervals

SECONDARY OUTCOMES:
operation time | During the procedure
  Evaluation of the operating time

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt